CLINICAL TRIAL: NCT01723319
Title: A Double Blind Randomized Controlled Evaluation of the HBLPADD-coil Transcranial Magnetic Stimulation (TMS) Device - Efficacy and Safety In Subjects With ADHD.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SH-0025-12
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: ADHD
Keywords: ADHD; TMS; brain stimulation; clinical improvement
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): deep TMS treatment
  Interventions: Device: HBLPADD coil deep TMS
- 2 (Sham Comparator): inactive treatment
  Interventions: Device: Sham

INTERVENTIONS:
Device: HBLPADD coil deep TMS — 20 daily deep TMS treatment
  Arms: 1
Device: Sham — inactive treatment
  Arms: 2

SUMMARY:
Objectives:The purpose of the study is to explore the efficacy and safety of HBLPADD Coil deep brain TMS in subjects with ADHD.

Patient Population: The intention is to treat 40 patients diagnosed with ADHD. The patients will be of all racial, ethnic and gender categories, ranging from 18 to 65 years of age.

Structure: The study is a randomized, prospective, 5 weeks, double blind study. Blinding: The treatment administrator and the study personnel and patients will be masked to the treatment being administrated.

The study group will receive active dTMS treatment and the control group will receive an inactive, sham treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18-65(male and female).
2. Diagnosed as suffering from Attention-Deficit Hyperactivity Disorder according to the DSM IV.
3. Patients taking medication for ADHD will give their consent to stop those medication 48 before entering the study and throughout the daily treatments.
4. Gave informed consent for participation in the study.
5. If referred by the treating psychiatrist, he or she approves of the subjects participation in the study.

Exclusion Criteria:

1. Suffering from other diagnosis on axis 1.
2. antipsychotic treatment with stabilizers; medications from the Benzodiazepines group are allowed, if need be,to a maximum dosage of 2 mg lorazepam.
3. History of lack of tolerance to TMS.
4. Axis 2 diagnosis according to the DSM IV.
5. Substantial suicidal risk as judged by the treating psychiatrist or by an independent psychiatrist.
6. Attempted suicide in the past year.
7. High and not controlled blood pressure.
8. History of epilepsy, seizure, or hot spasm.
9. History of epilepsy or seizure in first degree relatives.
10. History of a significant head injury
11. History of metal in the head (outside the mouth space).
12. Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
13. Use of hearing aids for hearing loss.
14. History of frequent or severe headaches.
15. History of drug or alcohol abuse during the last year.
16. Inability to achieve satisfying level of communication with the subject.
17. Participation in current clinical study or clinical study within 30 days prior to this study
18. Patients declared as legally incompetent, with an appointed physical guardian and/or cannot sign informed consent due to cognitive incompetence.
19. Women - Pregnancy or not using a reliable method of birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy will be examined by the change in the CAARS questionnaire from the baseline visit to the determination visit in the treatment group compared to the control group. | 5 weeks

SECONDARY OUTCOMES:
clinical improvement as measured using Clinical global Impression (CGI). | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: yechiel levkovitz, MD, Principal Investigator — Shalvata Mental Health Center
Locations (1):
- Shalvata, Hod HaSharon, Israel